CLINICAL TRIAL: NCT07072442
Title: Integrative Chinese and Western Medicine for Knee Osteoarthritis: Model of Patient Centered Healthcare and Shared Decision-making
Brief Title: Integrative Chinese and Western Medicine for Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NMRPG8Q6021
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthristis
MeSH Terms: interventions — Phytotherapy; Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Western medicine (Active Comparator): Western medicine treatment only
  Interventions: Drug: Western Medicine
- Herbal medicine and acupuncture (Experimental): Western medicine combined herbal medicine and acupuncture
  Interventions: Procedure: herbal medicine and acupuncture
- herbal medicine (Experimental): Western medicine combined herbal medicine
  Interventions: Drug: herbal medicine
- Acupuncture (Experimental): western medicine combined acupuncture
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Drug: Western Medicine — Western medicine treatment only
  Arms: Western medicine
Procedure: herbal medicine and acupuncture — Western medicine combined acupuncture and herbal medicine treatemnt
  Arms: Herbal medicine and acupuncture
Drug: herbal medicine — Western medicine combined herbal medicine
  Arms: herbal medicine
Procedure: acupuncture — western medicine combined acupuncture
  Arms: Acupuncture

SUMMARY:
This study aims to investigate if an integrated approach combining Traditional Chinese and Western medicine can better treat knee osteoarthritis. The goal is to see if this combined therapy can more effectively reduce pain severity and frequency, leading to an improved quality of life for KOA patients. Additionally, the study will explore the underlying mechanisms of pain and anti-inflammation related to KOA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged above 18 years old
* Kellgren-lawrence grading scale ≥ II
* Numerical rating scale (NRS) ≥ 4

Exclusion Criteria:

* History of bone tumor
* Pregnancy
* History of bilateral knee replacement
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
WOMAC | From enrollment to 3 months after treatment completion.
  Western Ontario and McMaster Universities Osteoarthritis (WOMAC) subscale
NRS | From enrollment to 3 months after treatment completion.
  Numerical rating scale (NRS) score for pain
Lequesne's index | From enrollment to 3 months after treatment completion.
  Lequesne's index

IPD SHARING:
Plan to Share IPD: No